# Pneumo-CLL study: Immunogenicity of the Currently Recommended Pneumococcal Vaccination Schedule in Patients with Chronic Lymphocytic Leukaemia.

Protocol Date: 01-06-2020

### **PROTOCOL**

Principal Investigator: K. de Heer

Co-investigator: H. Garcia Garrido

Writing committee: A. Goorhuis

H. Otten

H. Visser

F. de Boer

J. Droogendijk

I. Verpoorte

D. Issa

R. te Raa

R. van der Griend

H. van der Straaten

M-D. Levin

S. Kersting

A. Kater

#### 1. Introduction

Patients with chronic lymphocytic leukaemia (CLL) are at increased risk of both invasive pneumococcal disease (IPD) and community acquired pneumonia (CAP) caused by Streptococcus pneumoniae [1-3]. Therefore, international guidelines recommend pneumococcal vaccination for all CLL patients, preferably before initiation of treatment. The recommended vaccination schedule consists of Prevenar13®, a 13-valent pneumococcal conjugated vaccine (PCV13) followed 2 months later by Pneumovax23, a 23-valent polysaccharide vaccine (PPSV23) [4, 5].

The immunological efficacy of this sequential vaccination schedule in CLL patients is unknown. Previous studies have only investigated responses to either PCV13 or PPSV23 alone (Table 1) [6-15]. Responses to PPSV23 alone are poor in CLL patients [7, 9, 10, 14, 15]. Responses to the 7-valent pneumococcal conjugated vaccine (PCV7) or PCV13 are higher compared to responses to PPSV23, but lower compared to responses in healthy individuals [6, 8, 15]. More advanced disease stage and lower baseline IgG negatively influence responses to vaccination (Table 1) [6, 14, 15].

| Study | Year | N (final analysis) | Population | Vaccination schedule | Serologic respone definition | Response rate | Factors associated with response |
|---|---|---|---|---|---|---|---|
| A) Studies | investi | gating sch | nedules containing | conjugated vaccine | es (PCV7/PCV13) | | |
| Sinisalo et al<br>(8) | 2007 | 73 | n=49 CLL (15%<br>steroids, 22% chemo,<br>80% Binet A, median<br>disease duration 2<br>years); n=24 healthy | PCV7 only | ≥ 2 fold IgG rise AND serotype<br>specific IgG ≥ 0.35 mcg/l for at least<br>6/7 PCV7 serotypes | 24% CLL; 71% controls | Less advanced disease; no past or ongoing chemotherapy; normal IgG. |
| aiarski et al<br>6) | 2014 | 39 | Treatment naive CLL<br>(n=24); Healthy (n=15) | PCV13 only | ≥2 fold Total anti-pneumococcal IgG | 58.3% CLL; 100%<br>controls | Lower stage of CLL, higher total IgG |
| Andrick et al<br>(11) | 2017 | 8 | n=4 CLL + ibrutinib; n=<br>4 CLL - ibrutinib | PCV13 only | ≥2-fold increase in 3 or more out of 13 serotypes | Ibrutinib 0%;<br>No Ibrutinib 100% | x |
| Svensson et<br>al (15) | 2018 | 128 | Treatment naive CLL patients | PCV7 versus PPSV23<br>(RCT) | Serotype specific OPA titers to<br>PCV13 serotypes > Lowel Limit of<br>Quantification (OPA titers =<br>interpolated reciprocal serum<br>dilution resulting in complement-<br>mediated killing of 50% of the assay<br>bacteria) | PCV13: 32% ; PPSV23<br>21% | Less advanced disease; higher total I IgG |
| indström et<br>al (13) | 2018 | 24 | CLL, follow-up study<br>of Sinisalo 2007 | PCV7 5 years before | Serotype specific IgG ≥ 0.35 mcg/l (per serotype) | For individual<br>serotypes 29-71% of<br>the patients were still<br>protected | х |
| Lindström et<br>al (12) | 2019 | 28 | CLL (n=20); healthy<br>controls (n=8), follow-<br>up study of Sinisalo<br>2007 | • | Serotype specific IgG for all PCV7 serotypes AND PPSV23 serotype 5 and 7 | 10-15% | Healthy controls had higher responses to all serotypes |
| B) Studies | investi | gating PPS | SV23 only | | | | |
| Hartkamp et<br>al (14) | 2001 | 24 | 57% Rai 0-1; 28% prior<br>chemothrapy; median<br>disease duration >36<br>months | PPSV23 | Protection: 2/3 serotypes 20% above<br>cut-off based on reference adult<br>hyperimmune plasma pool;<br>Response: >2 fold increase +<br>protection (definition above) | Response: 22%<br>Protection: improved<br>from 38% to 50% after<br>vaccine; | Higher disease stage + lower<br>baseline IgG; prior chemotherapy<br>negatively impacted responses |
| Sinisalo et al<br>(7) | 2001 | 27 | n=14 Binet A, n=8<br>Binet B n=9 Binet C),<br>median disease<br>duration 3 years. | PPSV23 | A significant proportionate change in total anti-pneumcoccal IgG (no cut off value given) | 0% | х |
| van der<br>Velden et al<br>(9) | 2007 | 49 | CLL >50% RAI 0; 20% previous chemotherapy | PPSV23 (with or without ranitidine) | Response =>4 fold increase in IgG to<br>3 serotypes; Protection: ≥0,35<br>mcg/ml | Response: 1%<br>response;<br>'Protection' increased<br>from 45%-59% | Ranitidine did not generate better responses |
| Safdar et al<br>(10) | 2008 | 32 | 87% had previous<br>chemotehrapy and<br>73% anti-CD20 | PPSV23 (n=7); PPSV23<br>+ G-CSF injections<br>(n=25) | ≥2-fold IgG rise and level<br>>0.5mcg/ml for all 6 measured<br>seorypes | 0% (0-17% per<br>individual serotype) | G-CSF did not generate better responses |

## 2. Objective

The aim of this observational cohort study is to assess the immunogenicity of the currently recommended vaccination schedule of PCV13 followed by PPSV23 in CLL patients.

## 3. Study design

As part of routine care, all adult CLL patients naïve to pneumococcal vaccination and cared for in the participating centers receive one dose of Prevenar13® followed by one dose of Pneumovax23® 2 months later. According to the current local standard of care for immunosuppressed individuals, the response to vaccination is assessed by measuring pneumococcal antibody levels before and 4-8 weeks after vaccination [16, 17]. In this non-interventional cohort study we will ask informed consent to all vaccinated CLL patients to collect their clinical data and laboratory results for study purposes.

#### 4. Inclusion criteria

All adult CLL patients

- naïve to pneumococcal vaccination,
- having received one dose of Prevenar13®,
- followed by one dose of Pneumovax23® 2 months later,
- in whom pneumococcal antibody levels before and 4-8 weeks after vaccination are measured, and
- in whom a complete data collection is possible.

#### 5. Data collection

After we obtain informed consent clinical data will be collected according to a standardized electronic case report form (Castor EDC). Variables included in the case report form are:

- sex
- smoking behaviour
- age at the moment of the PCV vaccine administration
- comorbidities (charlson comorbitiy index)
- before vaccination (as determined in the 6 weeks prior to vaccination)
  - Rai stage (I/II/III)
  - past or ongoing chemotherapy
  - ongoing steroid treatment
  - past or ongoing therapy with a monoclonal anti-CD20 antibody (and date of last infusion)
  - total IgG level
  - lymphocyte count, haemoglobin and platelet level
- pre-vaccination pneumococcal IgG levels
- post-vaccination pneumococcal IgG levels
- date of PCV and PPSV23 vaccine administration
- date of antibody measurements

#### Laboratory methods and definitions

Serotype-specific pneumococcal immunoglobulin G (IgG) concentrations to 5 pneumococcal serotypes shared across both vaccines (6B, 9V, 14, 19F, 23F) and 4 serotypes unique to PPSV23 (8, 15B, 20, 33F) will be determined in the immunology laboratory of the UMC Utrecht. A validated multiplex immunoassay will be used (Luminex® technology). Serologic response will be defined as a ≥4-fold increase in serotype specific anti-pneumococcal IgG for ≥70% of measured. Serologic protection will be defined as an antibody concentration ≥1.3 mcg/ml for ≥70% of all measured serotypes, according to the definition of the *American Academy of Allergy, Asthma & Immunology* [18]. In addition, because most previous studies (Table 1) used the WHO cut-off for protection in infants (≥0.35 mcg/ml) we will also analyse our data by the infant correlate of protection to be able to compare our results with previous studies [19].

## 6. Data Analysis

The primary outcome of the study is serologic response rate (SRR) after vaccination. Secondary outcomes of interest are serologic protection rates (SPR) after vaccination analysed by the 2 most widely accepted serologic cut-offs described above, geometric mean antibody concentrations before and after vaccination, and factors associated with response to vaccination, such as age, treatment status and disease stage. To this end, we will perform a multivariable logistic regression analysis, starting with all previously mentioned clinical variables of interest and using a stepwise backward selection method based on p-value <0.1. For data analysis, we will use IBM SPSS version 24.0 (Chicago, Illinois) software. We will apply an  $\alpha$  significance level of 0.05. Means and standard deviations will be presented for normally distributed data, and medians and interquartile ranges for non-normally distributed data. The  $\chi 2$  test will be used for dichotomous variables and the Student t test or Mann-Whitney U test for normally or non-normally distributed continuous variables, respectively. The Wilcoxon signed-rank test will be used to compare median pre- and post-vaccination antibody concentrations.

## 7. Ethical considerations and privacy

For this non-interventional study, participants are not exposed to additional study procedures. Vaccination and assessment of vaccination responses are according to local standard of care. A waiver for medical ethical assessment has been issued by the Medical Ethical Committee of the Amsterdam UMC-Location AMC. Informed consent will be asked of each individual patient for use of their data for research purposes. A data protection impact analysis will be performed in collaboration with privacy advisors of all participating hospitals.

#### 8. References

1. Backhaus, E., et al., *Epidemiology of invasive pneumococcal infections: manifestations, incidence and case fatality rate correlated to age, gender and risk factors.* BMC Infect Dis, 2016. **16**: p. 367.

Protocol Date: 01-06-2020

- 2. Williams, A.M., et al., *Analysis of the risk of infection in patients with chronic lymphocytic leukemia in the era of novel therapies*. Leuk Lymphoma, 2018. **59**(3): p. 625-632.
- 3. Lindstrom, V., et al., *Invasive pneumococcal disease in patients with haematological malignancies before routine use of conjugate vaccines in Finland.* Infect Dis (Lond), 2016. **48**(5): p. 399-402.
- 4. Mikulska, M., et al., *Vaccination of patients with haematological malignancies who did not have transplantations: guidelines from the 2017 European Conference on Infections in Leukaemia (ECIL 7)*. Lancet Infect Dis, 2019. **19**(6): p. e188-e199.
- 5. Rubin, L.G., et al., 2013 IDSA clinical practice guideline for vaccination of the immunocompromised host. Clin Infect Dis, 2014. **58**(3): p. 309-18.
- 6. Pasiarski, M., et al., *Antibody and plasmablast response to 13-valent pneumococcal conjugate vaccine in chronic lymphocytic leukemia patients--preliminary report.* PLoS One, 2014. **9**(12): p. e114966.
- 7. Sinisalo, M., et al., Response to vaccination against different types of antigens in patients with chronic lymphocytic leukaemia. Br J Haematol, 2001. **114**(1): p. 107-10.
- 8. Sinisalo, M., et al., *Antibody response to 7-valent conjugated pneumococcal vaccine in patients with chronic lymphocytic leukaemia.* Vaccine, 2007. **26**(1): p. 82-7.
- 9. Van der Velden, A.M., et al., *The effect of ranitidine on antibody responses to polysaccharide vaccines in patients with B-cell chronic lymphocytic leukaemia*. Eur J Haematol, 2007. **79**(1): p. 47-52.
- 10. Safdar, A., et al., Multiple-dose granulocyte-macrophage-colony-stimulating factor plus 23-valent polysaccharide pneumococcal vaccine in patients with chronic lymphocytic leukemia: a prospective, randomized trial of safety and immunogenicity. Cancer, 2008. **113**(2): p. 383-7.
- 11. Andrick, B., et al., *Lack of adequate pneumococcal vaccination response in chronic lymphocytic leukaemia patients receiving ibrutinib.* Br J Haematol, 2018. **182**(5): p. 712-714.
- 12. Lindstrom, V., et al., *Antibody response to the 23-valent pneumococcal polysaccharide vaccine after conjugate vaccine in patients with chronic lymphocytic leukemia*. Hum Vaccin Immunother, 2019. **15**(12): p. 2910-2913.
- 13. Lindstrom, V., et al., *Antibody persistence after pneumococcal conjugate vaccination in patients with chronic lymphocytic leukemia*. Hum Vaccin Immunother, 2018. **14**(6): p. 1471-1474.
- 14. Hartkamp, A., et al., *Antibody responses to pneumococcal and haemophilus vaccinations in patients with B-cell chronic lymphocytic leukaemia*. Vaccine, 2001. **19**(13-14): p. 1671-7.
- 15. Svensson, T., et al., *Pneumococcal conjugate vaccine triggers a better immune response than pneumococcal polysaccharide vaccine in patients with chronic lymphocytic leukemia A randomized study by the Swedish CLL group.* Vaccine, 2018. **36**(25): p. 3701-3707.
- 16. AMC. http://www2.hematologie-amc.nl/MATCH-RVP-009\_revaccinatie 2018.
- 17. RIVM, Landelijke adviezen voor vaccinatie bij chronisch inflammatoire aandoeningen. 2018.
- 18. Orange, J.S., et al., *Use and interpretation of diagnostic vaccination in primary immunodeficiency: a working group report of the Basic and Clinical Immunology Interest Section of the American Academy of Allergy, Asthma & Immunology.* J Allergy Clin Immunol, 2012. **130**(3 Suppl): p. S1-24.
- 19. Jodar, L., et al., Serological criteria for evaluation and licensure of new pneumococcal conjugate vaccine formulations for use in infants. Vaccine, 2003. **21**(23): p. 3265-72.